CLINICAL TRIAL: NCT03132467
Title: A Pilot Pre-Surgical Study Evaluating Anti-PD-L1 Antibody (Durvalumab [MEDI4736]) Plus Anti-CTLA-4 Antibody (Tremelimumab) in Patients With Hormone Receptor Positive, HER2 Negative Breast Cancer
Brief Title: Durvalumab and Tremelimumab Before Surgery in Treating Patients With Hormone Receptor Positive, HER2 Negative Stage II-III Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0902; NCI-2018-01189 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0902 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-04-25; First posted 2017-04-27 (Actual); Results first posted 2022-02-17 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Estrogen Receptor Positive; HER2/Neu Negative; Progesterone Receptor Positive; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: interventions — durvalumab; Immunoglobulin G; Disulfides; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tremelimumab, durvalumab) (Experimental): Patients receive tremelimumab IV over 1 hour and durvalumab IV over 1 hour on day 1. Treatment repeats every 4 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo a biopsy and receive standard of care neoadjuvant chemotherapy before undergoing surgery.
  Interventions: Biological: Durvalumab; Biological: Tremelimumab

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Biological: Tremelimumab — Given IV
  Other Names: Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP-675; CP-675,206; CP-675206; Ticilimumab

SUMMARY:
This early phase I trial studies the side effects of durvalumab and tremelimumab before surgery in treating patients with hormone receptor positive, HER2 negative stage II-III breast cancer. Immunotherapy with monoclonal antibodies, such as durvalumab and tremelimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility of enrolling patients with hormone receptor positive (HR+)/human epidermal growth factor receptor negative (HER2-) breast cancer onto a trial evaluating investigational agents prior to initiating standard neoadjuvant chemotherapy.

II. To evaluate the safety and tolerability of tremelimumab plus durvalumab in patients with HR+/HER2- breast cancer.

SECONDARY OBJECTIVES:

I. To assess immunologic/molecular responses to tremelimumab and durvalumab in patients with HR+/HER2- breast cancer who receive the combination therapy.

EXPLORATORY OBJECTIVES:

I. To evaluate the pathologic response in patients with HR+/HER2- breast cancer receiving tremelimumab plus durvalumab prior to initiating standard neoadjuvant chemotherapy.

OUTLINE:

Patients receive tremelimumab intravenously (IV) over 1 hour and durvalumab IV over 1 hour on day 1. Treatment repeats every 4 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo a biopsy and receive standard of care neoadjuvant chemotherapy before undergoing surgery.

After completion of study treatment, patients are followed up until the time of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and any locally-required authorization (e.g., Health Insurance Portability and Accountability Act [HIPAA]) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Hormone receptor positive (defined as estrogen receptor [ER] and/or progesterone receptor [PR] positive), HER2 negative breast cancer that is clinically staged II-III with no known metastatic disease. ER and/or PR defined as positive if expression > 10% by immunohistochemistry (IHC). HER2 negative or non-amplified as determined by the current American Society of Clinical Oncology-College of American Pathologists (ASCO-CAP) criteria which are as follows: HER2 testing by immunohistochemistry (IHC) as 0 or 1+. If HER2 is 2+, ISH (in situ hybridization) must be performed. HER2 is positive if: IHC 3+ based on circumferential membrane staining that is complete, intense ISH positive based on: 1) Single-probe average HER2 copy number >= 6.0 signals/cell, 2) Dual-probe HER2/CEP17 ratio >= 2.0; c,e with an average HER2 copy number >= 4.0 signals/cell, 3) Dual-probe HER2/CEP17 ratio >= 2.0; c,e with an average HER2 copy number < 4.0 signals/cell, 4) Dual-probe HER2/CEP17 ratio < 2.0; c,e with an average HER2 copy number >= 6.0 signals/cell
* Chemotherapy is planned for the patient in the neoadjuvant setting
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count (ANC) >=1.5 x 10^9/L (>= 1500 per mm^3)
* Platelet count >= 100 x 10^9/L (>= 100,000 per mm^3)
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only upon treating physician, principal investigators (PI) or co-PIs approval
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be =< 5 x ULN
* Creatinine clearance (CL) > 40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance
* Female subjects must either be of non-reproductive potential (i.e., post-menopausal by history: >= 60 years old and no menses for >= 1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative urine pregnancy test upon study entry
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
* Participation in another clinical study with an investigational product during the last 1 month prior to initiation of therapy
* Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab or an anti-CTLA4, including tremelimumab
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease >= 5 years before the first dose of study drug and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease e.g., cervical cancer in situ
* Has received therapy for this current diagnosis of breast cancer including endocrine therapy or chemotherapy
* A single QT interval corrected for heart rate (QTc) >= 470 ms. If an electrocardiogram (ECG) is interpreted to be a prolonged QT interval, 2 additional ECGs will be obtained and the PI will then evaluate all three ECGs and determine whether the patient should be excluded. Mean QT interval corrected for heart rate (QTc) >= 470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's correction
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab or tremelimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Active or prior documented autoimmune disease within the past 2 years

  * NOTE: Subjects with vitiligo, Graves disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* History of primary immunodeficiency
* History of allogeneic organ transplant
* History of hypersensitivity to durvalumab or tremelimumab or any excipient
* History of hypersensitivity to the combination or comparator agent (if applicable)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Known history of previous clinical diagnosis of tuberculosis
* History of leptomeningeal carcinomatosis
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab or tremelimumab
* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Subjects with uncontrolled seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2024-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer K Litton, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a feasibility trial of combined checkpoint blockade in patients with HR+/HER2 neg primary breast cancer to determine whether the strategy of combined checkpoint blockade therapy prior to chemotherapy could be an effective frontline therapy. Patients were eligible if they had hormone receptor positive, HER2 negative breast cancer and had neoadjuvant chemotherapy planned.
Pre-assignment Details: 16 participants enrolled, 8 participants were inevaluable.
Groups:
- Treatment (Tremelimumab, Durvalumab): Patients were treated with durvalumab at a dose of 1500 mg and tremelimumab at a dose of 75 mg, both administered IV, for 2 cycles on days 1 and 28 Patients then received standard neoadjuvant chemotherapy prior to breast surgery Pre- and post-treatment tumor biopsies and blood samples were available for 5 out of 8 patients and were analyzed by CyTOF, IHC, and NanoString"
Period: Overall Study
Arm/Group | Treatment (Tremelimumab, Durvalumab)
Started | 8
Completed | 4
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Tremelimumab, Durvalumab)
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 55 [47 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Enrolling 15 Patients Within 2 Years
Description: Feasibility established if all 15 patients enroll within 12 months of starting the study. The start date for measuring feasibility will be the date the first patient is screened.
Time Frame: Up to 2 years
Population: The trials primary endpoint of 15 participants enrollment feasibility within 2 years was NOT met due to early termination of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tremelimumab, Durvalumab)
Number analyzed (Participants) | 8
Participants | 8

2. Primary Outcome: Safety and Tolerability of Tremelimumab Plus Durvalumab in Participants With HR+/HER2 Neg Breast Cancer.
Description: To evaluate the safety and tolerability of tremelimumab plus durvalumab in patients with HR+/HER2 neg breast cancer. Adverse events per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event [CTCAE] v4.03.
Time Frame: 2 months
Measure: Number; unit: adverse events
Groups:
- Treatment (Tremelimumab, Durvalumab): Participants with stage II or III HR+/HER2 negative breast cancer who were to receive neoadjuvant chemotherapy
Arm/Group | Treatment (Tremelimumab, Durvalumab)
Number analyzed (Participants) | 8
adverse events
  Serious Adverse Events | 3
  Adverse Events | 8

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Treatment (Tremelimumab, Durvalumab)
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tremelimumab, Durvalumab) (N=8)
Colitis (Gastrointestinal disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tremelimumab, Durvalumab) (N=8)
Conjunctivits (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 1 (1)
Hot flashes (Endocrine disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The trial was stopped early after 2 of 8 patients experienced G3 immunerelated adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT03132467/Prot_SAP_000.pdf